CLINICAL TRIAL: NCT00703911
Title: A Prospective Observational Registry on the Use of NovoSeven® (Activated Recombinant Human Factor VIIa) for on Demand Treatment of Mild to Moderate Bleeds in Haemophilia A and B Patients With Inhibitors
Brief Title: Observational Registry of NovoSeven® Used as On-demand Treatment of Bleeds in Patients With Haemophilia A and B With Inhibitors
Acronym: ONE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: F7HAEM-3507
Record Dates: First submitted 2008-06-19; First posted 2008-06-24 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A With Inhibitors; Haemophilia B With Inhibitors
MeSH Terms: interventions — Factor VII

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- activated recombinant human factor VII: Male patients above 2 years of age with haemophilia A or B who have developed inhibitors and have been prescribed on-demand treatment of activated recombinant human factor VII at any dose for treatment of mild to moderate spontaneous bleeds
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Treatment of patients experiencing bleeds at the discretion of the physician/caregiver
  Other Names: activated recombinant human factor VII

SUMMARY:
This study was conducted in Africa, Europe, the Middle-East and South America. The primary objective of this registry was to observe the use of single dose and multi-dose use of activated recombinant human factor VII and to compare short-term outcomes, including effectiveness, safety, quality of life and treatment satisfaction with the approved treatments.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with haemophilia A or B with inhibitors
* Experience mild to moderate spontaneous bleeds which require on-demand treatment and who are currently prescribed activated recombinant human factor VII
* Be able and willing to provide informed consent (or proxy consent by caregiver, if applicable), as required by local research ethics committee, governmental or regulatory authorities
* Be willing to provide information on at least one alternate contact person in the event that the patient be somehow lost-to-follow-up over the course of registry participation (not applicable if patient is withdrawn)

Exclusion Criteria:

* Known hypersensitivity to the active substance or the excipients in the formulation of activated recombinant human factor VII, or to mouse, hamster or bovine protein

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with haemophilia A or B with inhibitors, using activated recombinant human factor VII as on-demand treatment
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2008-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- Novo Nordisk Investigational Site, Algiers, Algeria
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Brussels, Belgium
- Novo Nordisk Investigational Site, Prague, Czechia
- Novo Nordisk Investigational Site, Paris La Défense Cedex, France
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Rome, Italy
- Novo Nordisk Investigational Site, Alphen aan den Rijn, Netherlands
- Novo Nordisk Investigational Site, Warsaw, Poland
- Novo Nordisk Investigational Site, Paço de Arcos, Portugal
- Novo Nordisk Investigational Site, Riyadh, Saudi Arabia
- Novo Nordisk Investigational Site, Sandton, South Africa
- Novo Nordisk Investigational Site, Malmo, Sweden
- Novo Nordisk Investigational Site, Istanbul, Turkey (Türkiye)
- Novo Nordisk Investigational Site, Crawley, United Kingdom
- Novo Nordisk Investigational Site, Caracas, Venezuela

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activated Recombinant Human Factor VII
Started | 102
Completed | 92
Not Completed | 10
Not completed — Death | 1
Not completed — Physician Decision | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.3 (16.37)
Age, Customized [Number; unit: participants]
  2 - 12 years | 35
  above 12 - 17 years | 14
  18 years or above | 53
Gender [Count of Participants; unit: Participants]
  Female | 0
  Male | 102
Region of Enrollment [Number; unit: participants]
  Algeria | 17
  Austria | 3
  Belgium | 4
  Czech Republic | 1
  France | 16
  Germany | 4
  Italy | 16
  Netherlands | 1
  Poland | 9
  Portugal | 1
  Saudi Arabia | 2
  South Africa | 8
  Sweden | 1
  Turkey | 6
  United Kingdom | 7
  Venezuela | 6
Peak inhibitor titre [Number; unit: participants]
  At least 5 Bethesda Units | 91
  Less than 5 Bethesda Units | 11
Outcome of immune tolerance induction (ITI) treatment [Number; unit: participants]
  None | 66
  Unsuccessful | 20
  Successful, with inhibitor recurrence | 5
  Ongoing ITI | 11
Estimated number of bleeds for the 6 months preceding enrolment in registry [Number; unit: participants]
  None | 9
  1 - 6 (1 or less per month) | 65
  6 - 12 (1 - 2 per month) | 13
  12 - 18 (2 - 3 per month) | 12
  18 (more than 3 per month) | 2
  Data missing | 1
Primary treatment pattern for the 6 months preceding enrolment in registry [Number; unit: participants]
  On-demand | 88
  Prophylaxis | 13
  Data missing | 1
Primary treatment type and dose for the 6 months preceding enrolment in registry [Number; unit: participants]
  Multiple dose 90 mcg/kg NovoSeven® | 44
  Single dose 270 mcg/kg NovoSeven® | 28
  Other dose regimen NovoSeven® | 17
  Other bypassing agent (e.g., FEIBA) | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Bleed Treatments Resulting in Effective Bleed Resolution (All Bleed Episodes)
Description: The percentage of bleed treatments successfully resulting in bleed resolution. Analysis only considers the patient's opinion of effectiveness at 9 hours, with a rating of "Effective" considered as successful treatment.
Time Frame: within 9 hours of first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose, n=494 | 61.7
  Low initial dose, n=156 | 67.9
  Intermediate initial dose, n=127 | 62.2
  High initial dose, n=211 | 56.9

2. Primary Outcome: Percentage of Bleed Treatments Resulting in Effective Bleed Resolution (Spontaneous Bleed Episodes)
Description: as for outcome 1
Time Frame: within 9 hours of first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose, n=324 | 59.0
  Low initial dose, n=92 | 62.6
  Intermediate initial dose, n=91 | 60.4
  High initial dose, n=141 | 55.7

3. Primary Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief (All Bleed Episodes)
Description: The percentage of participants with effective pain relief. Pain relief was a subjective assessment made by the patient during treatment of a bleed episode.
Time Frame: within 9 hours of first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose, n=494 | 71.3
  Low initial dose, n=156 | 82.1
  Intermediate initial dose, n=127 | 60.6
  High initial dose, n=211 | 69.7

4. Primary Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief (Spontaneous Bleed Episodes)
Description: as for outcome 3
Time Frame: within 9 hours of first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose, n=324 | 68.0
  Low initial dose, n=92 | 79.1
  Intermediate initial dose, n=91 | 58.2
  High initial dose, n=141 | 67.1

5. Secondary Outcome: Percentage of Bleed Treatments Resulting in Effective Haemostasis (Cessation of Bleeds) by Time Point (All Bleed Episodes)
Description: Effective haemostasis at 3 different time points for all bleeds. Patient reported outcomes are reported over 1 hour, 3 hours and 6 hours.
Time Frame: 1 hour, 3 hours and 6 hours, respectively, after first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose (1 hour), n=494 | 21.1
  Low initial dose (1 hour), n=156 | 16.8
  Intermediate initial dose (1 hr), n=127 | 25.8
  High initial dose (1 hour), n=211 | 21.5
  Any initial dose (3 hours), n=494 | 36.9
  Low initial dose (3 hours), n=156 | 32.5
  Intermediate initial dose (3 hrs), n=127 | 41.1
  High initial dose (3 hours), n=211 | 37.6
  Any initial dose (6 hours), n=494 | 50.8
  Low initial dose (6 hours), n=156 | 51.3
  Intermediate initial dose (6 hrs), n=127 | 51.2
  High initial dose (6 hours), n=211 | 50.2

6. Secondary Outcome: Percentage of Bleed Treatments Resulting in Effective Haemostasis (Cessation of Bleeds) by Time Point (Spontaneous Bleed Episodes)
Description: as for outcome 5
Time Frame: 1 hour, 3 hours and 6 hours, respectively, after first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose (1 hour), n=324 | 19.3
  Low initial dose (1 hour), n=92 | 7.7
  Intermediate initial dose (1 hr), n=91 | 24.4
  High initial dose (1 hour), n=141 | 23.6
  Any initial dose (3 hours), n=324 | 36.9
  Low initial dose (3 hours), n=92 | 27.8
  Intermediate initial dose (3 hrs), n=91 | 40.7
  High initial dose (3 hours), n=141 | 40.3
  Any initial dose (6 hours), n=324 | 48.1
  Low initial dose (6 hours), n=92 | 43.3
  Intermediate initial dose (6 hrs), n=91 | 50.5
  High initial dose (6 hours), n=141 | 49.6

7. Secondary Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief by Time Point (All Bleed Episodes)
Description: Effective pain relief at 3 different time points for all bleeds. Patient reported outcomes are reported over 1 hour, 3 hours and 6 hours.
Time Frame: 1 hour, 3 hours and 6 hours, respectively, after first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose (1 hour), n=494 | 27.7
  Low initial dose (1 hour), n=156 | 29.9
  Intermediate initial dose (1 hr), n=127 | 19.8
  High initial dose (1 hour), n=211 | 30.8
  Any initial dose (3 hours), n=494 | 53.1
  Low initial dose (3 hours), n=156 | 59.7
  Intermediate initial dose (3 hrs), n=127 | 47.2
  High initial dose (3 hours), n=211 | 51.7
  Any initial dose (6 hours), n=494 | 66.0
  Low initial dose (6 hours), n=156 | 77.8
  Intermediate initial dose (6 hrs), n=127 | 57.7
  High initial dose (6 hours), n=211 | 62.3

8. Secondary Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief by Time Point (Spontaneous Bleed Episodes)
Description: Effective pain relief at 3 different time points for spontaneous bleeds. Patient reported outcomes are reported over 1 hour, 3 hours and 6 hours.
Time Frame: 1 hour, 3 hours and 6 hours, respectively, after first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any initial dose (1 hour), n=324 | 24.7
  Low initial dose (1 hour), n=92 | 24.4
  Intermediate initial dose (1 hr), n=91 | 18.7
  High initial dose (1 hour), n=141 | 28.8
  Any initial dose (3 hours), n=324 | 49.1
  Low initial dose (3 hours), n=92 | 55.6
  Intermediate initial dose (3 hrs), n=91 | 44.0
  High initial dose (3 hours), n=141 | 48.2
  Any initial dose (6 hours), n=324 | 62.8
  Low initial dose (6 hours), n=92 | 77.5
  Intermediate initial dose (6 hrs), n=91 | 55.6
  High initial dose (6 hours), n=141 | 58.0

9. Secondary Outcome: Total Number of Injections (All Bleed Episodes)
Description: The median number of injections required to treat individual bleed episodes.
Time Frame: individual bleed episode
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Median (Inter-Quartile Range); unit: injections
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
injections
  Any initial dose, n=494 | 2 [1 to 3]
  Low dose, n=156 | 2 [2 to 3]
  Intermediate dose, n=127 | 2 [1 to 3]
  High dose, n=211 | 1 [1 to 2]

10. Secondary Outcome: Total Number of Injections (Spontaneous Bleed Episodes)
Description: The median number of injections required to treat individual bleed episodes.
Time Frame: individual bleed episode
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Median (Inter-Quartile Range); unit: injections
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
injections
  Any initial dose, n=324 | 2 [1 to 3]
  Low dose, n=92 | 2 [2 to 3]
  Intermediate dose, n=91 | 2 [1 to 3]
  High dose, n=141 | 1 [1 to 2]

11. Secondary Outcome: Total Exposure (Cumulative Dose) to Activated Recombinant Human Factor VII (All Bleed Episodes)
Description: The median total cumulative dose required to treat individual bleed episodes.
Time Frame: individual bleed episode
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level. Excludes bleeds episodes with greater than 24 hours between 1st and 2nd rFVII dose where total cumulative dose recorded likely reflects treatment of re-bleeding or prophylactic/maintenance dosing
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
mcg/kg
  Any initial dose, n=494 | 270 [43 to 2160]
  Low dose, n=156 | 267 [43 to 1632]
  Intermediate dose, n=127 | 256 [123 to 2160]
  High dose, n=211 | 270 [250 to 1822]

12. Secondary Outcome: Total Exposure (Cumulative Dose) to Activated Recombinant Human Factor VII (Spontaneous Bleed Episodes)
Description: The median total cumulative dose required to treat individual bleed episodes.
Time Frame: individual bleed episode
Population: Analysis set is spontaneous bleed episodes. Excludes bleeds episodes with > 24 hours between 1st and 2nd rFVII dose where total cumulative dose recorded likely reflects treatment of re-bleeding or prophylactic/maintenance dosing, and 2 bleed episodes categorised as CNS that would not meet criteria of mild to moderate spontaneous bleed episodes
Measure: Median (Full Range); unit: mcg/kg
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
mcg/kg
  Any initial dose, n=324 | 184 [90 to 1632]
  Low dose, n=92 | 284 [123 to 2160]
  Intermediate dose, n=91 | 270 [250 to 1822]
  High dose, n=141 | 270 [90 to 2160]

13. Secondary Outcome: Percentage of Patients Reporting Satisfaction With Symptom Relief (All Bleed Episodes)
Description: Patient rate of satisfaction with symptom relief for the bleed episode overall on a 7-point Likert scale. Completion of questionnaire was voluntary. A Likert scale is an ordered, multiple choice questionnaire from which respondents choose one option that best aligns with their view of the particular outcome being measured. Scale answers ranged from extremely satisfied to extremely dissatisfied. The percentage of bleed episodes for which patients reported "extremely satisfied", "very satisfied" or "satisfied" is presented.
Time Frame: duration of bleed episode
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any dose, n=494 | 72.7
  Low dose, n=156 | 82.1
  Intermediate dose, n=127 | 69.3
  High dose, n=211 | 67.8

14. Secondary Outcome: Percentage of Bleed Treatments Resulting in Patient Satisfaction With Symptom Relief (Spontaneous Bleed Episodes)
Description: as for outcome 13
Time Frame: duration of bleed episode
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any dose, n=324 | 68.2
  Low dose, n=92 | 75.0
  Intermediate dose, n=91 | 69.2
  High dose, n=141 | 63.1

15. Secondary Outcome: Percentage of Bleed Treatments Resulting in Patient Satisfaction With Ease of Use (All Bleed Episodes)
Description: Rate of ease of use related to activated recombinant human factor VII on a 7-point Likert scale. Completion of questionnaire was voluntary. A Likert scale is an ordered, multiple choice questionnaire from which respondents choose one option that best aligns with their view of the particular outcome being measured. Scale answers ranged from extremely difficult to extremely easy. The percentage of bleed episodes for which patients reported "extremely easy", "very easy" or "easy" is presented.
Time Frame: duration of bleed episode
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any dose, n=494 | 74.9
  Low dose, n=156 | 84.6
  Intermediate dose, n=127 | 74.8
  High dose, n=211 | 67.8

16. Secondary Outcome: Percentage of Bleed Treatments Resulting in Patient Satisfaction With Ease of Use (Spontaneous Bleed Episodes)
Description: as for outcome 15
Time Frame: duration of bleed episode
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any dose, n=324 | 69.1
  Low dose, n=92 | 81.5
  Intermediate dose, n=91 | 69.2
  High dose, n=141 | 61.0

17. Secondary Outcome: Overall Time to Cessation of Bleed/Achievement of Haemostasis (All Bleed Episodes)
Description: Median time to achievement of haemostasis/bleed cessation calculated using Kaplan Meier life table methods. If approximately 50% or less of bleeds achieved the endpoint in a given initial dose subgroup, the median cannot be calculated and it is reported as not applicable
Time Frame: duration of bleed episode
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
minutes
  Any dose, n=494 | 1200 [720 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing
  Low dose, n=156 | 720 [540 to 1430]
  Intermediate dose, n=127 | NA [NA to NA] — Since 50% or less of bleeds achieved the endpoint in the intermediate dose subgroup, the median cannot be calculated and it is reported as "not applicable" (NA)
  High dose, n=211 | 1200 [660 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing

18. Secondary Outcome: Overall Time to Cessation of Bleed/Achievement of Haemostasis (Spontaneous Bleed Episodes)
Description: as for outcome 17
Time Frame: duration of bleed episode
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
minutes
  Any dose, n=324 | 1200 [600 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing
  Low dose, n=92 | 600 [540 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing
  Intermediate dose, n=91 | NA [NA to NA] — Since 50% or less of bleeds achieved the endpoint in the intermediate dose subgroup, the median cannot be calculated and it is reported as "not applicable" (NA)
  High dose, n=141 | 1200 [540 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing

19. Secondary Outcome: Overall Time to Cessation/Achievement of Haemostasis (Spontaneous Bleed Episodes)
Description: as for outcome 17
Time Frame: duration of bleed episode
Population: Analysis set is spontaneous bleed episodes treated with any initial dose, excluding bleed episodes treated with more than one dose for which > 24 hours between the 1st and 2nd dose was reported (bleed episodes with > 24 hours between 1st and 2nd rFVIIa dose likely reflects treatment of re-bleeding or prophylactic/maintenance dosing)
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
minutes
  Any dose, n=270 | 600 [480 to 780]
  Low dose, n=87 | 600 [540 to NA] — Using Kaplan-Meier methods to calculate the median time to event takes into account the censoring of data at the upper part of the distribution. If the upper limit falls to the right of the censoring time, then it will be missing
  Intermediate dose, n=80 | NA [NA to NA] — Since 50% or less of bleeds achieved the endpoint in the intermediate dose subgroup, the median cannot be calculated and it is reported as "not applicable" (NA)
  High dose, n=103 | 480 [330 to 720]

20. Secondary Outcome: Childrens' Health Related Quality of Life (Haemo-QoL): Overall Score
Description: The Haemo-QoL is a specific multidimensional validated and reliable questionnaire used to assess quality of life in patients with haemophilia. Scores are reported on a 0 to 100 scale-higher scores indicate more impairment.
Time Frame: Baseline (week 0) and and registry discontinuation (up to 28 months)
Population: A subset of paediatric subjects age 4 to 16 (inclusive) included in the study that completed the questionnaire at baseline and/or at discontinuation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 7
scores on a scale
  Baseline, n=7 | 47.49 (11.08)
  Discontinuation, n=7 | 54.12 (10.19)

21. Secondary Outcome: Adults' Health Related Quality of Life (Haemo-QoL-A): Overall Score
Description: The adult Haemo-QoL-A is a specific multidimensional validated and reliable questionnaire used to assess quality of life in patients with haemophilia. Scores are reported on a 0 to 100 scale-higher scores indicate more impairment.
Time Frame: Baseline (week 0) and and registry discontinuation (up to 28 months)
Population: A subset of adult subjects above 16 years included in the study that completed the questionnaire at baseline and/or at discontinuation
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 11
scores on a scale
  Baseline, n=11 | 35.31 (9.69)
  Discontinuation, n=10 | 34.46 (12.14)

22. Other Pre Specified Outcome: Percentage of Bleed Treatments Resulting in Effective Haemostasis (Cessation of Bleed) by Dose Level (All Bleed Episodes)
Description: Percentage of bleeds with effective haemostasis within 9 hours of first injection of activated recombinant human factor VII. Patient reported assessments were sorted into 3 sub-categories: "effective" = bleed resolved or substantially improved; "partially effective" = bleed with some improvement; "ineffective" = bleed with no change or with worsening.
Time Frame: within 9 hours after first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any, effective | 61.7
  Any, partially effective | 26.7
  Any, ineffective | 11.7
  Low, effective | 67.5
  Low, partially effective | 21.2
  Low, ineffective | 11.3
  Intermediate, effective | 62.1
  Intermediate, partially effective | 31.5
  Intermediate, ineffective | 6.5
  High, effective | 57.1
  High, partially effective | 27.8
  High, ineffective | 15.1

23. Other Pre Specified Outcome: Percentage of Bleed Treatments Resulting in Effective Haemostasis (Cessation of Bleed) by Dose Level (Spontaneous Bleed Episodes)
Description: as for outcome 22
Time Frame: within 9 hours after first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any, effective | 59.0
  Any, partially effective | 29.3
  Any, ineffective | 11.7
  Low, effective | 62.1
  Low, partially effective | 21.8
  Low, ineffective | 16.1
  Intermediate, effective | 60.4
  Intermediate, partially effective | 36.3
  Intermediate, ineffective | 3.3
  High, effective | 56.1
  High, partially effective | 29.5
  High, ineffective | 14.4

24. Other Pre Specified Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief by Initial Dose (All Bleed Episodes)
Description: Percentage of bleeds with effective pain relief within 9 hours of first injection of activated recombinant human factor VII. Patient reported assessments were sorted into 3 sub-categories: "Better" = pain resolved or decreased substantially; "Same" = no change; "Worsened" = pain worsening.
Time Frame: within 9 hours after first injection
Population: Analysis set is all bleed episodes, regardless of bleed type or initial dose level
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any, better | 71.3
  Any, same | 25.6
  Any, worsened | 3.1
  Low, better | 60.0
  Low, same | 39.2
  Low, worsened | 0.8
  Intermediate, better | 82.4
  Intermediate, same | 15.0
  Intermediate, worsened | 2.6
  High, better | 69.9
  High, same | 25.2
  High, worsened | 4.9

25. Other Pre Specified Outcome: Percentage of Bleed Treatments Resulting in Effective Pain Relief by Initial Dose (Spontaneous Bleed Episodes)
Description: as for outcome 24
Time Frame: within 9 hours after first injection
Population: Analysis set is spontaneous bleed episodes treated with any initial dose
Measure: Number; unit: percentage of bleed episodes
Arm/Group | Activated Recombinant Human Factor VII
Number analyzed (Participants) | 85
percentage of bleed episodes
  Any, better | 68.1
  Any, same | 28.7
  Any, worsened | 3.2
  Low, better | 79.8
  Low, same | 16.9
  Low, worsened | 3.4
  Intermediate, better | 58.2
  Intermediate, same | 40.7
  Intermediate, worsened | 1.1
  High, better | 67.2
  High, same | 28.5
  High, worsened | 4.4

ADVERSE EVENTS:
Arm/Group | Activated Recombinant Human Factor VII
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to Novo Nordisk for review at least 60 days before submission for publication or presentation. The investigator will recognize the integrity of a multi-centre study by not publishing data derived from the individual site until the combined results from the completed registry have been published in full, or the sponsor confirms there will be no multi-centre registry publication.